CLINICAL TRIAL: NCT02617745
Title: Impact of the Platelet Level During Radiotherapy Associated With Temozolomide in Patients Treated for Glioblastoma
Brief Title: Impact of the Platelet Level in Patients Treated for Glioblastoma With Temozolomid
Acronym: GLIOPLAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB 15.02
Record Dates: First submitted 2015-11-16; First posted 2015-12-01 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: Stupp protocol, glioblastoma, thrombocytopenia
MeSH Terms: conditions — Glioblastoma; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stupp protocol (Experimental): Blood assessment of the platelet level every week during the radiotherapy phase and every cycle during the chemotherapy
  Interventions: Other: Platelet level determination

INTERVENTIONS:
Other: Platelet level determination — evaluate the predictive value of a biological test performed in the radio-chemotherapy phase in patients suffering from glioblastoma. For this the platelet level will be determined each wek during the radiotherapy phase and each cycle during the chemotherapy phase

SUMMARY:
The purpose of GLIOPLAK is to evaluate the predictive value of a biological test performed in the radio-chemotherapy phase in patients suffering from glioblastoma. The studied parameter is the variation in platelet count during the radio-chemotherapy phase. The main objective is to identify early in Stupp protocol a group of patients having high risk to undergo thrombocytopenia in maintenance phase of temozolomide. With this result an algorithm of platelet monitoring for patients treated with Stupp protocol wil be proposed.

DETAILED DESCRIPTION:
Glioblastoma is the most common primitive cerebral tumor. Currently its optimal treatment is based on a multidisciplinary approach combining an initial surgical resection, if feasible, then Stupp protocol. Stupp protocol consists of two phases: first phase involves external radiotherapy with concomitant oral temozolomide at a dose of 75mg/m2 per day for about six weeks. After 4 weeks of therapy break, maintenance phase begins with temozolomide alone, for a period of 6 cycles (1 cycle = 5 days over 28). The dose of temozolomide is 150mg/m2 on the first cycle followed by 200 mg/m2. One major limiting toxicity of temozolomide is hematologic, especially thrombocytopenia. They occur in around 15 and 20% of patients in maintenance phase. Thrombocytopenia has an impact on the schedule of Stupp protocol such as dose reduction or even early discontinuation. Currently no predictive marker of thrombocytopenia in the maintenance phase was identified. Such marker could be of major interest to adapt biological and clinical follow-up by patient in maintenance phase. We conduct a retrospective analysis on a cohort of patients suffering from glioblastoma and treated with Stupp protocol. We found that a decrease in platelet count during the radio-chemotherapy phase could be highly predictive of protocol changes in maintenance phase of temozolomide due to thrombocytopenia. The main objective of GLIOPLAK is to prospectively confirm the predictive value of this test and to evaluate the prognostic impact of the occurrence of thrombocytopenia <100,000/mm3. Secondary objective of GLIOPLAK are to describe all limiting toxicities in maintenance phase, to constitute a prospective biological collection and to collect biological samples to perform pharmacological analysis (pharmacogenomics and pharmacokinetics parameters).

ELIGIBILITY:
Inclusion Criteria:

* Age Superior to 18 years
* Inform consent form signed
* Newly diagnosed (histologically) glioblastoma
* Stupp protocol treatment
* with social insurance

Exclusion Criteria:

* Not inform consent form signed
* participation to another clinical trial
* other cancer
* background of hematological pathology
* patient under guardianship, curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Number of time where platelet level was Under 100 000 per mm3 | one year and 6 months
  Determination of platelet level to predict the risk of thrombocytopenia

SECONDARY OUTCOMES:
Overall survival | 3 years
  time between inclusion and death
Therapeutic modifications | one year and 6 months
  Proportion of patient with treatment modifications

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Di Fiore, MD, PhD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

REFERENCES:
- [Derived] Fontanilles M, Heisbourg JD, Daban A, Di Fiore F, Pepin LF, Marguet F, Langlois O, Alexandru C, Tennevet I, Ducatez F, Pilon C, Plichet T, Mokbel D, Lesueur C, Bekri S, Tebani A. Metabolic remodeling in glioblastoma: a longitudinal multi-omics study. Acta Neuropathol Commun. 2024 Oct 12;12(1):162. doi: 10.1186/s40478-024-01861-5. PMID 39394177
- [Derived] Daban A, Beaussire-Trouvay L, Leveque E, Alexandru C, Tennevet I, Langlois O, Veresezan O, Marguet F, Clatot F, Di Fiore F, Sarafan-Vasseur N, Fontanilles M. Prognostic value of circulating short-length DNA fragments in unresected glioblastoma patients. Transl Oncol. 2024 Apr;42:101897. doi: 10.1016/j.tranon.2024.101897. Epub 2024 Feb 9. PMID 38340682
- [Derived] Fontanilles M, Marguet F, Beaussire L, Magne N, Pepin LF, Alexandru C, Tennevet I, Hanzen C, Langlois O, Jardin F, Laquerriere A, Sarafan-Vasseur N, Di Fiore F, Clatot F. Cell-free DNA and circulating TERT promoter mutation for disease monitoring in newly-diagnosed glioblastoma. Acta Neuropathol Commun. 2020 Nov 4;8(1):179. doi: 10.1186/s40478-020-01057-7. PMID 33148330